CLINICAL TRIAL: NCT02762578
Title: A Trial Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart and BIAsp 30 in Subjects With Type 2 Diabetes BOOST: INTENSIFY PREMIX/ALL 2
Brief Title: Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart and BIAsp 30 in Subjects With Type 2 Diabetes
Acronym: BOOST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3598; 2011-000085-36 (EudraCT Number); U1111-1118-8578 (Other: WHO); CTR20150689 (Other: Chinese FDA)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp BID (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- BIAsp 30 BID (Active Comparator)
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Twice daily subcutaneous (sc, under the skin) injection.
  Arms: IDegAsp BID
Drug: biphasic insulin aspart — Twice daily subcutaneous (sc, under the skin) injection.
  Arms: BIAsp 30 BID

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare efficacy and safety of insulin degludec/insulin aspart and BIAsp 30 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female at least 18 years of age
* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Insulin treated subjects on current treatment: basal insulin, premixed insulin or a self-mixed insulin regimen, all administered once daily (OD) or BID with or without metformin. The treatment regimen should have remained unchanged for at least 8 weeks prior to randomisation
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* Body mass index (BMI) equal or below 40.0 kg/m^2

Exclusion Criteria:

* Treatment with sulphonylureas, meglitinides, DPP-4 inhibitors, alpha-glycosidase inhibitors within 8 weeks prior to screening (Visit 1) or thiazolidinediones (TZDs) or GLP-1 receptor agonists within 12 weeks prior to screening (Visit 1)
* Anticipated change in concomitant medication known to interfere significantly with glucose metabolism, such as systemic corticosteroids, beta-blockers and monoamine oxidase (MAO) inhibitors
* Anticipated significant lifestyle changes during the trial according to the discretion of the investigator, e.g. shift work (including permanent night/evening shift workers), as well as highly variable eating habits
* Cardiovascular disease, within the last 6 months prior to screening (Visit 1), defined as: stroke; decompensated heart failure NYHA1 class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Any clinically significant disease or disorder, except for conditions associated with type 2 diabetes, which in the investigator's opinion could interfere with the results of the trial
* Previous participation in this trial. Participation is defined as screened.
* Known or suspected hypersensitivity to trial products or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (21):
- China (21):
  - Novo Nordisk Investigational Site, Hefei, Anhui
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Nanning, Guangxi
  - Novo Nordisk Investigational Site, Cangzhou, Hubei
  - Novo Nordisk Investigational Site, Baotou, Inner Mongolia
  - Novo Nordisk Investigational Site, Changzhou, Jiangsu
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Suzhou, Jiangsu
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Siping, Jilin
  - Novo Nordisk Investigational Site, Jinan, Shandong
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Chengdu, Sichuan
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
  - Novo Nordisk Investigational Site, Kunming, Yunnan
  - Novo Nordisk Investigational Site, Tianjin

REFERENCES:
- [Result] Yang W, Ma J, Hong T, Liu M, Miao H, Peng Y, Wang C, Xu X, Yang T, Nielsen AM, Pan L, Liu W, Zhao W. Efficacy and safety of insulin degludec/insulin aspart versus biphasic insulin aspart 30 in Chinese adults with type 2 diabetes: A phase III, open-label, 2:1 randomized, treat-to-target trial. Diabetes Obes Metab. 2019 Jul;21(7):1652-1660. doi: 10.1111/dom.13703. Epub 2019 Apr 4. PMID 30869183
- [Derived] Luo Q, Zhou L, Zhou N, Hu M. Cost-effectiveness of insulin degludec/insulin aspart versus biphasic insulin aspart in Chinese population with type 2 diabetes. Front Public Health. 2022 Oct 18;10:1016937. doi: 10.3389/fpubh.2022.1016937. eCollection 2022. PMID 36330105
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 sites were approved for recruiting subjects, of which 40 sites screened and randomized the subjects.
Pre-assignment Details: Insulin treated subjects on current treatment: basal insulin, premixed insulin or a self-mixed insulin regimen, all administered once daily or twice daily (BID) with or without metformin. The treatment regimen should have remained unchanged for at least 8 weeks prior to randomisation.
Groups:
- IDegAsp BID: Subjects received subcutaneous (s.c.) injections of insulin degludec/insulin aspart (IDegAsp) twice daily (BID) for 26 weeks. Subjects started insulin treatment at dose corresponding to their pre-trial insulin treatment. The insulin dose adjustments aimed to reach pre-breakfast and pre-dinner self-measured plasma glucose (SMPG) ≤ 5.0 mmol/L, based on the subject's pre-breakfast and pre-dinner SMPG. The dose taken with main evening meal was adjusted according to mean pre-breakfast plasma glucose measured on the day of adjustment and the two preceding days. The dose taken at breakfast was adjusted according to mean pre-main evening meal plasma glucose measured on the three days preceding the adjustment day. If one of the PG values was below target (< 4.0 mmol/L), the corresponding dose was to be reduced. If one or more SMPG values were missing, the adjustment was to be performed on remaining SMPG values. Subjects continued the pre-trial treatment with metformin at stable dose.
- BIAsp 30 BID: Subjects received s.c. injections of biphasic insulin aspart 30 (BIAsp 30, a mixture of soluble insulin aspart [IAsp] 30% and protaminated IAsp 70%) BID for 26 weeks. Subjects started insulin treatment at dose corresponding to their pre-trial insulin treatment. The insulin dose adjustments aimed to reach pre-breakfast and pre-dinner SMPG ≤5.0 mmol/L, based on the subject's pre-breakfast and pre-dinner SMPG. The dose taken with main evening meal was adjusted according to mean pre-breakfast plasma glucose measured on day of adjustment and the two preceding days. The dose taken at breakfast was adjusted according to mean pre-main evening meal plasma glucose measured on the three days preceding the adjustment day. If one of the PG values was below target (< 4.0 mmol/L), the corresponding dose was to be reduced. If one or more SMPG values were missing, the adjustment was to be performed on the remaining SMPG values. Subjects continued the pre-trial treatment with metformin at stable dose.
Period: Overall Study
Arm/Group | IDegAsp BID | BIAsp 30 BID
Started | 361 | 182
Exposed | 360 | 181
Completed | 346 | 172
Not Completed | 15 | 10
Not completed — Adverse Event | 1 | 6
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Unclassified | 6 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp BID | BIAsp 30 BID | Total
Number analyzed (Participants) | 361 | 182 | 543
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.64 (9.04) | 58.78 (9.41) | 59.35 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 83 | 246
  Male | 198 | 99 | 297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 361 | 182 | 543
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 361 | 182 | 543
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.32 (0.76) | 8.33 (0.77) | 8.32 (0.76)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] — Population: Number of participants analysed=participants with available data for FPG at baseline
  mmol/L
    number analyzed (Participants) | 355 | 180 | 535
    (all) | 9.07 (2.21) | 9.07 (2.49) | 9.07 (2.31)
Body weight [Mean (Standard Deviation); unit: kg] | 68.50 (11.63) | 69.41 (12.38) | 68.80 (11.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (%) (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c after 26 weeks of treatment. The response and change from baseline in response after 26 weeks are analysed using an analysis of covariance model with treatment, anti-diabetic therapy at screening and sex as fixed factors, age and baseline response as covariate. Missing values imputed using last observed value.
Time Frame: At 26 weeks
Population: Full analysis set. Number of subject analysed=subjects with available data for HbA1c
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 359 | 182
percentage of HbA1c | -1.48 (0.05) | -1.40 (0.06)
Statistical Analysis 1: Comparison: IDegAsp BID vs BIAsp 30 BID; Change from baseline in HbA1c after 26 weeks of treatments was analysed using an ANCOVA method with treatment, anti-diabetic therapy at screening and sex as fixed factors, and age and baseline HbA1c as covariates; Test type: Non-Inferiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 1: Primary analysis: Non-inferiority with respect to change from baseline in HbA1c (%) to week 26 for IDegAsp vs. BIAsp 30. Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval was below or equal to 0.4%; p = 0.2430, ANCOVA — Two-sided p-value for testing difference; Treatment contrast = -0.08, 95% CI 2-sided [-0.20 to 0.05]
Statistical Analysis 2: Comparison: IDegAsp BID vs BIAsp 30 BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — If non-inferiority was confirmed, the superiority of the IDegAsp group over the BIAsp 30 group was to be investigated. Superiority was considered confirmed if the upper bound of the two-sided 95% confidence interval, which was calculated using the FAS, was below 0%; p = 0.2430, ANCOVA — Two-sided p-value for testing difference; Treatment contrast = -0.08, 95% CI 2-sided [-0.20 to 0.05]

2. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose)
Description: Change from baseline in FPG at week 26. The response and change from baseline in response after 26 weeks are analysed using an analysis of covariance model with treatment, anti-diabetic therapy at screening and sex as fixed factors, age and baseline response as covariate. Missing values imputed using last observed value.
Time Frame: At 26 weeks
Population: Full analysis set. Number of subject analysed=subjects with available data for FPG.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 354 | 180
mmol/L | -2.99 (0.09) | -1.57 (0.13)
Statistical Analysis 1: Comparison: IDegAsp BID vs BIAsp 30 BID; Change from baseline in FPG after 26 weeks of treatment was analysed using an ANCOVA method with treatment, anti-diabetic therapy at screening and sex as fixed factors, and age and baseline FPG as covariates; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 2: Superiority with respect to change from baseline in FPG to week 26 for IDegAsp vs. BIAsp 30 (Provided that non-inferiority was confirmed for the primary endpoint) Superiority was considered confirmed if the 95% CI for the treatment difference (IDegAsp group-BIAsp 30 group) was entirely below zero; p < 0.0001, ANCOVA — Two-sided p-value for testing difference; Treatment Contrast = -1.42, 95% CI 2-sided [-1.74 to -1.10]

3. Secondary Outcome: Number of Treatment Emergent Nocturnal Confirmed Hypoglycaemic Episodes
Description: The number of events was analysed using a negative binomial model with a log-link function and the logarithm of the exposure time (100 years) for which a hypoglycaemic episode is considered treatment emergent as offset. The model included treatment, anti-diabetic therapy at screening and sex as fixed factors, and age as covariate. Confirmed hypoglycaemia is defined as either severe episodes or episodes with plasma glucose < 3.1 mmol/L (56 mg/dL) with or without symptoms. The nocturnal period was defined as the period between 00:01 and 05:59 a.m. (both inclusive). A treatment emergent hypoglycaemic episode was defined as an episode that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: Weeks 0-26
Population: Full analysis set. Number of subjects analysed=subjects with data available for nocturnal confirmed hypoglycaemic episodes.
Measure: Number; unit: events per 100 patient years of exposure
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 359 | 181
events per 100 patient years of exposure | 31.18 | 58.55
Statistical Analysis 1: Comparison: IDegAsp BID vs BIAsp 30 BID; The number of events was analysed using a Negative Binomial Model with a log-link function and the logarithm of the exposure time (100 years) for which a hypoglycaemic episode is considered treatment emergent as offset. The model included treatment, anti-diabetic therapy at screening and sex as fixed factors, and age as covariate; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 3: Superiority with respect to nocturnal confirmed hypoglycaemic episodes for IDegAsp vs. BIAsp 30 (provided that superiority with respect to change from baseline in FPG to week 26 was confirmed for IDegAsp vs. BIAsp 30). Superiority was considered confirmed if the 95% CI for the rate ratio (IDegAsp group/BIAsp 30 group) was entirely below one; p = 0.0112, Negative binomial regression model; Treatment Ratio = 0.53, 95% CI 2-sided [0.33 to 0.87]

4. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes
Description: The number of events was analysed using a negative binomial model with a log-link function and the logarithm of the exposure time (100 years) for which a hypoglycaemic episode is considered treatment emergent as offset. The model included treatment, anti-diabetic therapy at screening and sex as fixed factors, and age as covariate. Confirmed hypoglycaemia was defined as either severe episodes or episodes with plasma glucose < 3.1 mmol/L (56 mg/dL) with or without symptoms. A treatment emergent hypoglycaemic episode was defined as an episode that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment.
Time Frame: Weeks 0-26
Population: Full analysis set. Number of subjects analysed=subjects with data available for confirmed hypoglycaemic episodes.
Measure: Number; unit: events per 100 patient years of exposure
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 359 | 181
events per 100 patient years of exposure | 223.56 | 394.17
Statistical Analysis 1: Comparison: IDegAsp BID vs BIAsp 30 BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 4: Superiority with respect to confirmed hypoglycaemic episodes for IDegAsp vs. BIAsp 30 (provided that superiority with respect to nocturnal confirmed hypoglycaemic episodes for IDegAsp vs. BIAsp 30 was confirmed). Superiority was considered confirmed if the 95% CI for the rate ratio (IDegAsp group/BIAsp 30 group) was entirely below one; p = 0.0002, Negative binomial regression model; Treatment Ratio = 0.57, 95% CI 2-sided [0.42 to 0.77]

5. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body week at week 26. The response and change from baseline in response after 26 weeks are analysed using an ANCOVA model with treatment, anti-diabetic therapy at screening and sex as fixed factors, age and baseline response as covariate. Missing values imputed using last observed value.
Time Frame: Week 0, Week 26
Population: Full analysis set. Number of subject analysed=subjects with data available for body weight.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 359 | 182
kg | 2.82 (0.14) | 2.21 (0.19)
Statistical Analysis 1: Comparison: IDegAsp BID vs BIAsp 30 BID; The response and change from baseline in response after 26 weeks were analysed using an ANCOVA model with treatment, anti-diabetic therapy at screening and sex as fixed factors, age and baseline response as covariate; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 5: Superiority with respect to change from baseline in body weight for IDegAsp vs. BIAsp 30 (provided that Superiority with respect to confirmed hypoglycaemic episodes for IDegAsp vs. BIAsp 30 was confirmed). Superiority was considered confirmed if the 95% CI for the treatment difference (IDegAsp group-BIAsp 30 group) was entirely below zero; p = 0.0092, ANCOVA; Two-sided p-value for testing difference; Treatment contrast = 0.61, 95% CI 2-sided [0.15 to 1.08]

6. Secondary Outcome: Responder Without Confirmed Hypoglycaemic Episodes HbA1c Below 7.0%
Description: A responder for HbA1c without confirmed hypoglycaemia was defined as a subject who meets the HbA1c target (<7.0%) at end of trial without treatment emergent confirmed hypoglycaemia during the last 12 weeks of treatment or within 7 days after the last randomised treatment. Confirmed hypoglycaemia was defined as either severe episodes or episodes with plasma glucose < 3.1 mmol/L (56 mg/dL) with or without symptoms. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Missing data is imputed using last observed value.
Time Frame: At 26 weeks
Population: Full analysis set. Number of subjects analysed=subjects who have been exposed for at least 12 treatment weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 348 | 173
Participants
  Yes | 153 | 48
  No | 195 | 125
Statistical Analysis 1: Comparison: IDegAsp BID vs BIAsp 30 BID; The endpoint was analysed in a logistic regression model using a logit link, including treatment, sex and anti-diabetic treatment at screening as fixed effects, and age and HbA1c as covariates; Test type: Superiority — Stepwise hierarchical testing procedure was applied for confirmatory endpoints: Step 6: Superiority with respect to subjects achieving HbA1c < 7% at end of trial without confirmed hypoglycaemia for IDegAsp vs. BIAsp 30 (provided that superiority with respect to change from baseline in body weight was confirmed). Superiority was considered confirmed if the 95% CI for the odds ratio (IDegAsp group/BIAsp 30 group) was entirely above one; p = 0.0002, Regression, Logistic — Two-sided p-value for testing difference; Treatment Ratio = 2.22, 95% CI 2-sided [1.47 to 3.35]

7. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs)
Description: A treatment emergent adverse event was defined as an episode that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. Incidence of AEs was reported in terms of rate, defined as number of adverse events divided by patient years of exposure (PYE) multiplied by 100 (1 PYE=365.25 days).
Time Frame: Weeks 0-26
Population: Safety analysis set included all subjects receiving at least one dose of IDegAsp or BIAsp.
Measure: Number; unit: events per 100 PYE
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 360 | 181
events per 100 PYE | 321.74 | 348.82

8. Secondary Outcome: Responder for HbA1c (HbA1c <7%) After 26 Weeks of Treatment
Description: Number of subjects with HbA1c <7% after 26 weeks of treatment. Missing HbA1c data was imputed using last observed value.
Time Frame: Week 26
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 361 | 182
Participants
  Yes | 201 | 88
  No | 160 | 94

9. Secondary Outcome: Responder for HbA1c (HbA1c <=6.5%) After 26 Weeks of Treatment
Description: Number of subjects with HbA1c <=6.5% after 26 weeks of treatment. Missing HbA1c data was imputed using last observed value.
Time Frame: Week 26
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 361 | 182
Participants
  Yes | 106 | 54
  No | 255 | 128

10. Secondary Outcome: Responder for HbA1c (HbA1c <7%) Without Severe Hypoglycaemic Episodes
Description: A responder for HbA1c without severe hypoglycaemia was defined as a subject who meets the HbA1c target (<7%) at end of trial without severe treatment emergent hypoglycaemia during the last 12 weeks of treatment or within 7 days after the last randomised treatment. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Missing HbA1c data was imputed using last observed value.
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects who have been exposed for at least 12 treatment weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 348 | 173
Participants
  Yes | 197 | 84
  No | 151 | 89

11. Secondary Outcome: Responder for HbA1c (HbA1c ≤6.5%) Without Confirmed Hypoglycaemic Episodes
Description: A responder for HbA1c without confirmed hypoglycaemia was defined as a subject who meets the HbA1c target (≤6.5%) at end of trial without treatment emergent confirmed hypoglycaemia during the last 12 weeks of treatment or within 7 days after the last randomised treatment. Confirmed hypoglycaemia was defined as either severe episodes or episodes with plasma glucose < 3.1 mmol/L (56 mg/dL) with or without symptoms. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Missing data is imputed using last observed value.
Time Frame: At 26 weeks
Population: Full analysis set. Number of subjects analysed=subjects who have been exposed for at least 12 treatment weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 348 | 173
Participants
  Yes | 82 | 26
  No | 266 | 147

12. Secondary Outcome: Responder for HbA1c (HbA1c ≤6.5%) Without Severe Hypoglycaemic Episodes
Description: A responder for HbA1c without severe hypoglycaemia was defined as a subject who meets the HbA1c target (≤6.5%) at end of trial without severe treatment emergent hypoglycaemia during the last 12 weeks of treatment or within 7 days after the last randomised treatment. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Missing HbA1c data was imputed using last observed value.
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects who have been exposed for at least 12 treatment weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 348 | 173
Participants
  Yes | 105 | 50
  No | 243 | 123

13. Secondary Outcome: 9-point Profile (SMPG) After 26 Weeks of Treatment
Description: SMPG values were recorded at 9 time-points: before and after (90 min after the start of the meal) breakfast, lunch, main evening meal, before bedtime, at 4 am and before breakfast on the next day. Missing values were imputed using last observed value.
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects with SMPG values available at individual timepoints.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 361 | 182
mmol/L
  Before breakfast: number analyzed (Participants) | 360 | 182
  Before breakfast | 5.81 (1.29) | 6.81 (1.90)
  90 minutes after start of breakfast: number analyzed (Participants) | 350 | 174
  90 minutes after start of breakfast | 8.68 (2.81) | 9.56 (3.25)
  Before lunch: number analyzed (Participants) | 351 | 175
  Before lunch | 6.47 (2.39) | 6.65 (2.50)
  90 minutes after start of lunch: number analyzed (Participants) | 350 | 173
  90 minutes after start of lunch | 10.22 (3.06) | 10.52 (3.17)
  Before main evening meal: number analyzed (Participants) | 359 | 182
  Before main evening meal | 7.09 (2.35) | 7.97 (2.92)
  90 minutes after the start of main evening meal: number analyzed (Participants) | 350 | 173
  90 minutes after the start of main evening meal | 9.35 (3.04) | 8.96 (3.26)
  Before bedtime: number analyzed (Participants) | 353 | 172
  Before bedtime | 8.65 (3.00) | 8.12 (2.89)
  At 4:00 a.m.: number analyzed (Participants) | 346 | 170
  At 4:00 a.m. | 6.00 (1.93) | 6.78 (1.95)
  Before breakfast the following day: number analyzed (Participants) | 360 | 180
  Before breakfast the following day | 5.69 (1.49) | 6.87 (1.82)

14. Secondary Outcome: Mean of the 9-point Profile (SMPG) After 26 Weeks of Treatment
Description: SMPG values were recorded at 9 time-points: before and after (90 min after the start of the meal) breakfast, lunch, main evening meal, before bedtime, at 4 am and before breakfast on the next day. Missing values were imputed using last observed value. The mean of 9-point profile (SMPG) was defined as the area under the profile divided by the measurement time and was calculated using the trapezoidal method.
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects with available data for SMPG.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 360 | 182
mmol/L | 7.70 (1.60) | 8.11 (1.71)

15. Secondary Outcome: Fluctuation in the 9-point Profile (SMPG) After 26 Weeks of Treatment
Description: SMPG values were recorded at 9 time-points: before and after (90 min after the start of the meal) breakfast, lunch, main evening meal, before bedtime, at 4 am and before breakfast on the next day. Missing values were imputed using last observed value. Fluctuation in 9-point SMPG profile is the average absolute difference to the mean of the profile of the 9-point SMPG measurements accumulated over the profile.
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects with available data for SMPG.
Measure: Median (Full Range); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 360 | 182
mmol/L | 1.40 [0.08 to 4.90] | 1.43 [0.04 to 4.18]

16. Secondary Outcome: 9-point Profile (SMPG) - Prandial Plasma Glucose (PG) Increment After 26 Weeks of Treatment
Description: SMPG values were recorded at 9 time-points: before and after (90 min after the start of the meal) breakfast, lunch, main evening meal, before bedtime, at 4 am and before breakfast on the next day. Missing values were imputed using last observed value. Prandial PG increment for each meal was derived from the 9-point profile (SMPG) as the difference between PG values after meal (90 min) and before meal. The reported results are mean prandial PG increment overall meals (the mean of all available meal increments).
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects with SMPG values available before and after (90 min after the start of the meal) breakfast, lunch, main evening meal.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 359 | 182
mmol/L | 2.95 (2.10) | 2.60 (2.15)

17. Secondary Outcome: 2-point Profile (SMPG) Measurements Obtained Throughout the Trial for Dose Adjustment - Time From Randomisation (Measured in Weeks) to Achieve Titration Targets
Description: 2-point profiles (SMPG): pre-breakfast and pre-dinner (main evening meal) SMPGs were to be taken for titration/dose adjustments. The pre-specified titration targets were to achieve SMPG level <5 mmol/L (90 mg/dL) both before breakfast and before main evening meal. For each target, the time from randomisation to the date a subject achieves the titration target for the first time was derived (Kaplan-Meier method). Reported results are time to all titration target (pre-breakfast and pre-dinner) was met for the first time.
Time Frame: From randomization till achievement of titration target (up to week 26)
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: week
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 361 | 182
week | NA [24.0 to NA] — Median and upper bound of inter-quartile range could not be calculated as inadequate number of subjects achieved the pre-defined titration target at the end of trial. | NA [NA to NA] — Median and IQR could not be calculated as inadequate number of subjects achieved the pre-defined titration target at the end of trial

18. Secondary Outcome: 2-point Profile (SMPG) Measurements Obtained Throughout the Trial for Dose Adjustment - Within-subject Variability as Measured by Coefficient of Variance (CV)% After 26 Weeks of Treatment
Description: The logarithm transformed SMPG values available before breakfast and main evening meal were analysed separately as repeated measures in a linear mixed model with treatment, anti-diabetic therapy at screening and sex as fixed factors, age as covariate and subject as random factor. The model assumed independent within- and between-subject errors with variances depending on treatment. Within-subject variability as measured by CoV% for a treatment could be calculated from the corresponding residual variance.
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects who contributed to this analysis.
Measure: Number; unit: Coefficient of variation
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 180
Coefficient of variation
  Before breakfast | 17.26 | 17.19
  Before main evening meal | 22.45 | 22.96

19. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association (ADA) Definition During 26 Weeks of Treatment
Description: ADA classification of hypoglycaemia:
  1. Severe: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
  2. Asymptomatic: An episode not accompanied by typical symptoms of hypoglycaemia, but with a measured PG level ≤3.9 mmol/L.
  3. Documented symptomatic: An episode during which typical symptoms of hypoglycaemia are accompanied by a measured PG level ≤3.9 mmol/L.
  4. Relative: An episode during which the person with diabetes reports any of the typical symptoms of hypoglycaemia, and interprets those as indicative of hypoglycaemia, but with a measured PG level >3.9 mmol/L.
  5. Probable symptomatic: An episode during which symptoms of hypoglycaemia are not accompanied by a PG determination but that was presumably caused by a PG level ≤3.9 mmol/L.
  Number of treatment emergent hypoglycaemic episodes were reported in terms of rate, defined as number of events divided by PYE multiplied by 100 (1 PYE=365.25 days).
Time Frame: Week 0-26
Population: Safety analysis set.
Measure: Number; unit: hypoglycaemic episodes per 100 PYE
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 360 | 181
hypoglycaemic episodes per 100 PYE | 1699.53 | 1585.31

20. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes in the Maintenance Period
Description: Confirmed hypoglycaemia was defined as either severe episodes or episodes with plasma glucose < 3.1 mmol/L (56 mg/dL) with or without symptoms. Severe: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Maintenance period was defined as the period from week 16 to end of treatment, including 1 week follow-up.
  Number of treatment emergent hypoglycaemic episodes were reported in terms of rate, defined as number of events divided by PYE multiplied by 100 (1 PYE=365.25 days).
Time Frame: From week 16 to end of treatment (week 26) + 1 week follow-up
Population: Safety analysis set
Measure: Number; unit: hypoglycaemic episodes per 100 PYE
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 360 | 181
hypoglycaemic episodes per 100 PYE | 159.08 | 361.18

21. Secondary Outcome: Number of Treatment Emergent Nocturnal (00:01-05:59) Confirmed Hypoglycaemic Episodes in the Maintenance Period
Description: Confirmed hypoglycaemia was defined as either severe episodes or episodes with plasma glucose < 3.1 mmol/L (56 mg/dL) with or without symptoms. Severe hypoglycaemia: An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. The nocturnal period was defined as the period between 00:01 and 05:59 a.m. (both inclusive). Maintenance period was defined as the period from week 16 to end of treatment, including 1 week follow-up.
  Number of treatment emergent hypoglycaemic episodes were reported in terms of rate, defined as number of events divided by PYE multiplied by 100 (1 PYE=365.25 days).
Time Frame: From week 16 to end of treatment (week 26) + 1 week follow-up
Population: Safety analysis set
Measure: Number; unit: hypoglycaemic episodes per 100 PYE
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 360 | 181
hypoglycaemic episodes per 100 PYE | 19.20 | 38.60

22. Secondary Outcome: Change in Health Related Quality of Life Questionnaire (SF -36)
Description: Change from baseline in SF-36 at week 26. The questionnaire contains 36 items across 8 domains and 2 summary scores. Score range: 0 (worst score) to 100 (best score). Missing data was imputed using last observed value.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of subjects analysed=subjects with data available for individual component of SF-36 questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 361 | 182
units on a scale
  Physical Score: number analyzed (Participants) | 359 | 181
  Physical Score | 0.19 (6.89) | -0.13 (6.61)
  Physical Functioning: number analyzed (Participants) | 359 | 182
  Physical Functioning | -1.01 (6.85) | -0.50 (6.58)
  Role-Physical: number analyzed (Participants) | 359 | 181
  Role-Physical | 0.41 (8.88) | -0.18 (8.92)
  Bodily Pain: number analyzed (Participants) | 360 | 182
  Bodily Pain | 0.93 (10.10) | -0.71 (10.38)
  General Health: number analyzed (Participants) | 360 | 182
  General Health | 3.00 (10.24) | 2.19 (9.45)
  Mental Score: number analyzed (Participants) | 359 | 181
  Mental Score | 2.08 (9.65) | 0.72 (10.11)
  Vitality: number analyzed (Participants) | 360 | 182
  Vitality | 1.56 (9.57) | 0.69 (9.33)
  Social Functioning: number analyzed (Participants) | 360 | 182
  Social Functioning | 1.35 (8.46) | -0.12 (9.98)
  Role-Emotional: number analyzed (Participants) | 359 | 181
  Role-Emotional | 1.54 (10.60) | 1.01 (11.14)
  Mental Health: number analyzed (Participants) | 360 | 182
  Mental Health | 1.39 (9.53) | -0.17 (9.81)

23. Secondary Outcome: Change in Treatment Satisfaction Questionnaire (Treatment Related Impact Measure-diabetes [TRIM-D])
Description: Change from baseline in TRIM-D scores at week 26. TRIM-D score measured treatment satisfaction which included an overall score as well the subscale scores (daily life, diabetes management, compliance and psychological health). The scores were transformed to a 0-100 scale with higher scores indicating less treatment related impact. Missing data was imputed using last observed value.
Time Frame: Week 0, week 26
Population: Full analysis set. Number of subjects analysed=subjects with data available for TRIM-D total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 360 | 181
units on a scale | 4.87 (11.15) | 4.11 (10.49)

24. Secondary Outcome: Treatment Satisfaction Questionnaire (Treatment Related Impact Measures - Diabetes Device [TRIM-D Device])
Description: TRIM-D device is an eight item measure with two domains assessing Device Bother and Device Function. This captures information on the ease of use, convenience, and handling of the device(s) used to take diabetes medication. The measure has acceptable reliability, validity and ability to detect change. The scores were transformed to a 0-100 scale with higher scores indicating less treatment related impact. Missing data was imputed using last observed value.
Time Frame: At week 26
Population: Full analysis set. Number of subjects analysed=subjects with data available for TRIM-D device total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
units on a scale | 72.31 (14.78) | 69.43 (14.12)

25. Secondary Outcome: Device Specific Questionnaires I (How Easy or Difficult is it to Read the Dose Scale)
Description: Device Specific Questionnaires I (How easy or difficult is it to read the dose scale) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 220 | 104
  Fairly easy | 128 | 69
  Neither easy nor difficult | 10 | 5
  Rather difficult | 0 | 0

26. Secondary Outcome: Device Specific Questionnaires I (How Easy or Difficult do You Find it to Hold the Pen Stable When Injecting?)
Description: Device Specific Questionnaires I (How easy or difficult do you find it to hold the pen stable when injecting?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 228 | 99
  Fairly easy | 121 | 72
  Neither easy nor difficult | 8 | 7
  Very difficult | 1 | 0

27. Secondary Outcome: Device Specific Questionnaires I (How Easy or Difficult is it to Hear the Clicks for Each Unit Increment?)
Description: Device Specific Questionnaires I (How easy or difficult is it to hear the clicks for each unit increment?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 230 | 108
  Fairly easy | 119 | 63
  Neither easy nor difficult | 9 | 6
  Rather difficult | 0 | 1

28. Secondary Outcome: Device Specific Questionnaires I (How Easy or Difficult is it to Feel the Clicks for Each Unit Increment?)
Description: Device Specific Questionnaires I (How easy or difficult is it to feel the clicks for each unit increment?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 217 | 103
  Fairly easy | 128 | 65
  Neither easy nor difficult | 12 | 9
  Rather difficult | 1 | 1

29. Secondary Outcome: Device Specific Questionnaires I (How Easy or Difficult is it to Push Down the Injection Button?)
Description: Device Specific Questionnaires I (How easy or difficult is it to push down the injection button?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 224 | 89
  Fairly easy | 125 | 75
  Neither easy nor difficult | 9 | 14
  Rather difficult | 0 | 0

30. Secondary Outcome: Device Specific Questionnaires I (How Easy/Difficult is it to Turn the Dose Selector When Choosing the Right Dose?)
Description: Device Specific Questionnaires I (How easy/difficult is it to turn the dose selector when choosing the right dose?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 222 | 99
  Fairly easy | 128 | 72
  Neither easy nor difficult | 7 | 6
  Rather difficult | 1 | 0

31. Secondary Outcome: Device Specific Questionnaires I (How Easy/Difficult is it to Know if the Push Button Has Been Pushed Completely Down?)
Description: Device Specific Questionnaires I (How easy/difficult is it to know if the push button has been pushed completely down?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult or Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 213 | 92
  Fairly easy | 134 | 77
  Neither easy nor difficult | 11 | 9

32. Secondary Outcome: Device Specific Questionnaires I (How Easy or Difficult is it to See the Dose Scale When Injecting?)
Description: Device Specific Questionnaires I (How easy or difficult is it to see the dose scale when injecting?) was measured on following categories: Very confident, Very easy, Fairly easy, Neither easy nor difficult, Rather difficult, and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very confident | 1 | 0
  Very easy | 215 | 94
  Fairly easy | 126 | 78
  Neither easy nor difficult | 14 | 4
  Rather difficult | 2 | 2

33. Secondary Outcome: Device Specific Questionnaires I (How Confident Are You That You Set the Insulin Dose Correctly Every Time?)
Description: Device Specific Questionnaires I (How confident are you that you set the insulin dose correctly every time?) was measured on following categories: Very confident, Rather confident, Fairly confident, Not very confident and Not at all confident. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very confident | 209 | 85
  Fairly confident | 43 | 26
  Rather confident | 106 | 65
  Not very confident | 0 | 2

34. Secondary Outcome: Device Specific Questionnaires I (How Confident Are You That You Inject the Correct Amount of Insulin Every Time?)
Description: Device Specific Questionnaires I (How confident are you that you inject the correct amount of insulin every time?) was measured on following categories: Very confident, Rather confident, Fairly confident, Not very confident and Not at all confident. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very confident | 202 | 83
  Fairly confident | 52 | 28
  Rather confident | 104 | 67

35. Secondary Outcome: Device Specific Questionnaires I (Overall, How Confident Are You in Your Management of Your Daily Insulin Injections Using This Pen?)
Description: Device Specific Questionnaires I (Overall, how confident are you in your management of your daily insulin injections using this pen?) was measured on following categories: Very confident, Fairly confident, Rather confident, Not very confident and Not at all confident. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very confident | 197 | 82
  Fairly confident | 59 | 39
  Rather confident | 102 | 57

36. Secondary Outcome: Device Specific Questionnaires I (Overall, How Confident Are You in Controlling Your Blood Sugar Level Using This Pen?)
Description: Device Specific Questionnaires I (Overall, how confident are you in controlling your blood sugar level using this pen?) was measured on following categories: Very confident, Fairly confident, Rather confident, Not very confident and Not at all confident. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very confident | 180 | 71
  Fairly confident | 85 | 60
  Rather confident | 92 | 42
  Not very confident | 1 | 3

37. Secondary Outcome: Device Specific Questionnaires I (How Suitable is the Pen to Use in Public?)
Description: Device Specific Questionnaires I (How suitable is the pen to use in public?) was measured on following scale: Very suitable, Fairly suitable, Rather suitable, Not very suitable and Not at all suitable. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very suitable | 129 | 60
  Fairly suitable | 117 | 64
  Rather confident | 0 | 1
  Rather suitable | 94 | 35
  Not very suitable | 18 | 18

38. Secondary Outcome: Device Specific Questionnaires I (How Confident Are You That the Air Shot Has Been Done Correctly?)
Description: Device Specific Questionnaires I (How confident are you that the air shot has been done correctly?) was measured on following categories: Very confident, Fairly confident, Rather confident, Not very confident and Not at all confident. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very confident | 157 | 73
  Fairly confident | 85 | 55
  Rather confident | 109 | 47
  Not very confident | 7 | 3

39. Secondary Outcome: Device Specific Questionnaires I (How Convenient do You Find the Size of the Pen?)
Description: Device Specific Questionnaires I (How convenient do you find the size of the pen?) was measured on following categories: Very convenient, Fairly convenient, Rather convenient, Not very convenient and Not at all convenient. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very convenient | 143 | 63
  Fairly convenient | 109 | 69
  Rather convenient | 101 | 42
  Not very convenient | 5 | 4

40. Secondary Outcome: Device Specific Questionnaires I (How Comfortable do You Find the Handling of the Pen?)
Description: Device Specific Questionnaires I (How comfortable do you find the handling of the pen?) was measured on following categories: Very comfortable, Fairly comfortable, Rather comfortable, Not very comfortable and Not at all comfortable. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very comfortable | 146 | 66
  Fairly comfortable | 107 | 68
  Rather comfortable | 104 | 44
  Not very comfortable | 1 | 0

41. Secondary Outcome: Device Specific Questionnaires I (Did You Have Any Problems Using the Pen?)
Description: Participants were asked to report whether they had any problems using the pen. Number of participants reporting "yes" and "no" are presented. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 1.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Yes | 12 | 8
  No | 346 | 169

42. Secondary Outcome: Device Specific Questionnaires II (How Easy or Difficult Was it to Learn How to Use This Pen?)
Description: Device Specific Questionnaires II (How easy or difficult was it to learn how to use this pen?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 2.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 206 | 92
  Fairly easy | 145 | 79
  Neither easy nor difficult | 7 | 7

43. Secondary Outcome: Device Specific Questionnaires II (How Easy or Difficult is it to Distinguish Between Dialling up and Down?)
Description: Device Specific Questionnaires II (How easy or difficult is it to distinguish between dialling up and down?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 2.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 203 | 91
  Fairly easy | 144 | 81
  Neither easy nor difficult | 10 | 6
  Rather difficult | 1 | 0

44. Secondary Outcome: Device Specific Questionnaires II (How Easy or Difficult is it to Inject Your Usual Insulin Dose?)
Description: Device Specific Questionnaires II (How easy or difficult is it to inject your usual insulin dose?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 2.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 193 | 93
  Fairly easy | 154 | 81
  Neither easy nor difficult | 11 | 3
  Rather difficult | 0 | 1

45. Secondary Outcome: Device Specific Questionnaires II (How Easy/Difficult is it to Reach the Dose Button When Inject Your Insulin Dose?)
Description: Device Specific Questionnaires II (How easy/difficult is it to reach the dose button when inject your insulin dose?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult and Very difficult. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 2.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 193 | 90
  Fairly easy | 153 | 82
  Neither easy nor difficult | 11 | 6
  Rather difficult | 1 | 0

46. Secondary Outcome: Device Specific Questionnaires II (How Easy or Difficult is it to Inject Yourself in Different Places of the Body Using This Pen?)
Description: Device Specific Questionnaires II (How easy or difficult is it to inject yourself in different places of the body using this pen?) was measured on following categories: Very easy, Fairly easy, Neither easy nor difficult, Rather difficult, Very difficult and Not applicable. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 2.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Very easy | 167 | 77
  Fairly easy | 169 | 85
  Neither easy nor difficult | 20 | 16
  Rather difficult | 1 | 0
  Very difficult | 1 | 0

47. Secondary Outcome: Device Specific Questionnaires II (How Confident Are You That the Full Dose Has Been Delivered?)
Description: Device Specific Questionnaires II (How confident are you that the full dose has been delivered?) was measured on following categories: Very confident, Fairly confident, Fairly easy, Rather confident, Not very confident and Not at all confident. Reported results are number of participants reporting the individual category of the question at week 26. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 2.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Not at all confident | 1 | 0
  Very confident | 184 | 79
  Fairly confident | 54 | 42
  Fairly easy | 0 | 1
  Rather confident | 117 | 56
  Not very confident | 2 | 0

48. Secondary Outcome: Device Specific Questionnaires II (Would You Recommend the Pen?)
Description: Participants were asked the question "would you recommend the pen?" Number of participants reporting "yes" and "no" are presented. Missing data was imputed using last observed value.
Time Frame: week 26
Population: Full analysis set. Number of participants analysed=subjects with data available for Device specific questionnaire 2.
Measure: Count of Participants; unit: Participants
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 358 | 178
Participants
  Yes | 338 | 161
  No | 19 | 17

ADVERSE EVENTS:
Time Frame: Week 0 to week 26 (+ 1 week of follow-up)
Description: A treatment emergent adverse event was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. Summary is based on the safety analysis set.
Arm/Group | IDegAsp BID | BIAsp 30 BID
All-Cause Mortality (participants affected / at risk) | 0/360 | 0/181
Serious Adverse Events (participants affected / at risk) | 16/360 | 14/181
Other Adverse Events (participants affected / at risk) | 109/360 | 65/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=360) | BIAsp 30 BID (N=181)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dysbacteriosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 2 (3)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=360) | BIAsp 30 BID (N=181)
Diabetic retinopathy (Eye disorders) | 36 (37) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 76 (90) | 46 (52)
Viral upper respiratory tract infection (Infections and infestations) | 9 (10) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT02762578/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT02762578/SAP_001.pdf